CLINICAL TRIAL: NCT02356926
Title: Cross Checking to Reduce Adverse Events Resulting From Medical Errors in the Emergency Department
Brief Title: Cross Checking to Reduce Adverse Events in the Emergency Department
Acronym: Charmed
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI14017; CRC13074 (Other: AP-HP)
Record Dates: First submitted 2015-02-02; First posted 2015-02-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-06

CONDITIONS: Emergency Patients
Keywords: Adverse events; Medical errors; Emergency department; Cross checking
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Usual care and routine management
- Cross checking: Systematic cross checking between emergency physicians at 11:30, 14:00 and 16:30

SUMMARY:
Multicenter cluster randomized study to evaluate the reduction of the rate of severe medical errors with implementation of systematic cross checkings between emergency physician.

DETAILED DESCRIPTION:
The CHARMED study is a prospective, multicenter, cluster-randomized cross-over study in six EDs in France. Centers will be randomly assigned to use routine management or systematic cross checking in the first period, and will use the alternative strategy in the second period (Fig 1). Patients will be recruited in six centers in France

In both periods, from 9am to 5pm, a CRT will be present in the ED to collect variables on providers and patients.

In the control period, usual care and routine management will be provided. In the intervention group, systematic cross-checking will be implemented three times a day from 8:30am to 6:00pm between emergency physicians. The CRT will seek emergency physicians (EP) by pairs for crosschecking. Senior physicians will use peer crosschecking (i.e. crosschecker will also be an emergency senior physician). The CRT will assist the pairing. Each EP will prepare to present all his or her current patients. Patient presentation will be will be protocolised (see below), although usual presentation will be sought as this is the presentation method already in place for handover. The crosschecking will occur in the presence of the CRT and in the ED, in any medical office staff room, or cubicle available.

Each EP will then have to present the patients he is actually taking care of, with brief description of the case. After a case has been presented by the EP, the comments and advice of the crosschecker will be sought.

In accordance to national and international recommendations 1,2,15, the following definitions will be used:

Medical Error: Failure of a planned action to be completed as intended, or the use of a wrong plan to achieve an aim. The severity of an error will be classified using the National Coordinating Council on Medical Error and Reporting (NCCMERP) from A to I 16, as shown in table 2.

Adverse event (AE): An injury that might have resulted from medical care (or lack thereof).

Near Miss: A medical error that has the potential to cause an adverse event, but did not either by chance or after an intervention. A near miss is an error of severity B, C or D.

Preventable AE: An AE associated with an error. A preventable AE is a medical error of severity E, F, G, H or I.

Severe Medical Error (SME): preventable AE or a near miss. The primary objective is to assess whether the implementation of Systematic Cross Serious unexplained guideline violation (local or national), even in the absence of any documented injury, will be considered an AE. Checking in the ED will reduce the rate of severe medical errors. The primary endpoint is the rate of SME in the seven days following ED visits. As previously described, the subsequent adverse events might not clearly appear in the ED settings, hence is considered as a SME 8. Hospital or ED re-attendance within the next 7 days will be also considered as an adverse event.

Secondary endpoints include the followings:

* Rate of AE and preventable AE
* Rate of Near Miss
* Severity of SME
* Factors associated to SME:

  * Related to patient (age, chief complaint, comorbidities, triage level)
  * Related to physician (grade, experience, number of physician involved, handoff)
  * Related to the ED visit (Time of visit, daily occupancy, crowding, waiting time, length of stay, total number of emergency physicians)

ELIGIBILITY:
Inclusion Criteria:

* All patients that visit the ED during one of the two periods of recruitment, monday to friday between 8:30am and 4:30pm, will be screened for inclusion. We chose this time interval as they correspond to period that can be exposed to a cross checking, which will occur at 11:30 am, 2:00 pm and 4:30 pm.

Exclusion Criteria:

* Patients whose care is not provided by an EP (for example psychiatrist or maxillo-facial surgeon)
* Scheduled return attendance to the ED
* Low severity, defined by

  1. Triage level 5 on a 1 to 5 scale 13,14
  2. Patients referred to a "minor" or "fast track" unit
  3. Patients discharged home less than 1 hours after first contact with an EP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency patients
Sampling Method: Probability Sample
Enrollment: 1680 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events and preventable adverse events in the 7 days after admission to the emergency | 7 days
  Occurrence of SAEs or "near miss" in the 7 days after admission to the emergency, defined as:
  * Serious Adverse Event (SAE): A damage or injury that may be the result of a medical intervention, or lack thereof.
  * Or "near miss" medical error with the potential to cause damage that has been intercepted or who luckily did not reach the patient

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Freund, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Freund Y, Goulet H, Leblanc J, Bokobza J, Ray P, Maignan M, Guinemer S, Truchot J, Feral-Pierssens AL, Yordanov Y, Philippon AL, Rouff E, Bloom B, Cachanado M, Rousseau A, Simon T, Riou B. Effect of Systematic Physician Cross-checking on Reducing Adverse Events in the Emergency Department: The CHARMED Cluster Randomized Trial. JAMA Intern Med. 2018 Jun 1;178(6):812-819. doi: 10.1001/jamainternmed.2018.0607. PMID 29710111
- [Derived] Freund Y, Rousseau A, Berard L, Goulet H, Ray P, Bloom B, Simon T, Riou B. Cross-checking to reduce adverse events resulting from medical errors in the emergency department: study protocol of the CHARMED cluster randomized study. BMC Emerg Med. 2015 Sep 4;15:21. doi: 10.1186/s12873-015-0046-1. PMID 26340941